CLINICAL TRIAL: NCT01800838
Title: Silicon Phthalocyanine Pc4 for Photodynamic Therapy of Cutaneous T-cell Lymphoma: Single and Repeated Photoexposures
Brief Title: Silicon Phthalocyanine 4 and Photodynamic Therapy in Stage IA-IIA Cutaneous T-Cell Non-Hodgkin Lymphoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Kevin Cooper MD (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor-Investigator, Kevin Cooper MD, Department Chairman, Dermatology, Case Comprehensive Cancer Center
Organization: Case Comprehensive Cancer Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CASE2411; NCI-2013-00089 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 4130 (Other: Orphan Product grant number)
Record Dates: First submitted 2013-02-26; First posted 2013-02-28 (Estimated); Results first posted 2019-05-16 (Actual); Last update posted 2019-05-16 (Actual); Status verified 2019-05

CONDITIONS: Recurrent Cutaneous T-cell Non-Hodgkin Lymphoma; Recurrent Mycosis Fungoides/Sezary Syndrome; Stage I Cutaneous T-cell Non-Hodgkin Lymphoma; Stage IA Mycosis Fungoides/Sezary Syndrome; Stage IB Mycosis Fungoides/Sezary Syndrome; Stage II Cutaneous T-cell Non-Hodgkin Lymphoma; Stage IIA Mycosis Fungoides/Sezary Syndrome
MeSH Terms: conditions — Lymphoma, T-Cell, Cutaneous; Mycosis Fungoides; Sezary Syndrome | interventions — SUB1 protein, human; Photochemotherapy; 1-phenyl-3,3-dimethyltriazene

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (silicon phthalocyanine 4 and PDT) (Experimental): Patients receive silicon phthalocyanine 4 topically and then undergo PDT.
  Interventions: Drug: silicon phthalocyanine 4; Drug: photodynamic therapy; Other: pharmacological study; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: silicon phthalocyanine 4 — Given topically
  Other Names: Pc 4; Pc-4 (Silicone phthalocyanine)
Drug: photodynamic therapy — Undergo PDT
  Other Names: Light Infusion Therapy™; PDT; therapy, photodynamic
Other: pharmacological study — Correlative studies
  Other Names: pharmacological studies
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This phase I trial studies the side effects and best dose of silicon phthalocyanine 4 and photodynamic therapy in treating patients with stage IA-IIA cutaneous T-cell non-Hodgkin lymphoma. Photodynamic therapy (PDT) uses a drug, silicon phthalocyanine 4, that becomes active when it is exposed to a certain kind of light. When the drug is active, cancer cells are killed. This may be effective against cutaneous T-cell non-Hodgkin lymphoma.

Funding Source - FDA OOPD

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the safety and maximum tolerated dose (MTD) that can be utilized for a single treatment of Pc 4-PDT (silicon phthalocyanine 4 photo dynamic therapy) on subjects with mycosis fungoides (MF)/cutaneous T-cell lymphoma (CTCL) stage IA-IIA, by evaluating an accelerated dose escalation protocol consisting of a single exposure to PDT using topically-applied Pc 4 and visible light at a wavelength of 675 nm, followed by assessment of skin biopsies to analyze cellular and molecular changes induced by Pc 4-PDT. (Cohort I)

II. Determine safety and tolerability of repeated light (PDT) exposures after a single application of Pc 4 to a MF/CTCL plaque, using topically-applied Pc 4 and visible light at a wavelength of 675nm, followed by assessment of skin biopsies to analyze cellular and molecular changes induced by Pc 4-PDT. (Cohort II)

III. Identification of targets for assessment of efficacy to assist in planning for a Phase II study.

OUTLINE: This is a dose-escalation study.

Patients receive silicon phthalocyanine 4 topically and then undergo PDT.

After completion of study treatment, patients are followed up at 24 hours, 1 week, 2 weeks, and 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with early stage MF (CTCL stage IA-IIA)
* Has at least 2 evaluable plaques
* Has been off systemic therapies for at least 4 weeks
* Has been off topical therapies for at least 2 weeks
* Has been off phototherapies for at least 2 weeks
* All skin photo-types will be included
* Subjects must have the ability to understand and the willingness to sign a written informed consent form
* Women of child-bearing potential must agree to utilize a birth control which results in a failure rate of less that 1% per year during the study; accepted forms of birth control for this study include: injections such as Depo-Provera and Lunelle, implants such as Norplant, and intra-uterine devices
* Sexually active males must agree to use a medically acceptable form of birth control for the duration of the study and for at least 3 months after the last dose of the study medication; appropriate birth control methods are using a condom with a spermicide or surgical sterilization

Exclusion Criteria:

* Active history of photosensitivity (e.g. xeroderma pigmentosum, lupus erythematosus, porphyria, severe polymorphous light eruption, solar urticaria)
* Any medical condition that could be aggravated or may cause extreme discomfort during the study period
* Lesions only on the face, scalp or other sites that would make biopsies not cosmetically acceptable
* Women of childbearing potential who are pregnant or attempting to become pregnant are excluded from this study
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to silicon phthalocyanine (Pc 4) or other agents used in this study
* Patients with uncontrolled intercurrent illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2013-04; Primary Completion 2014-09 (Actual); Study Completion 2015-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elma Baron, MD, Principal Investigator — University Hospitals Cleveland Medical Center, University Hospitals Seidman Cancer Center, Case Comprehensive Cancer Center
Locations (1):
- University Hospitals Cleveland Medical Center, University Hospitals Seidman Cancer Center, Case Comprehensive Cancer Center, Cleveland, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study recruited patients between April 2013 and April 2015 at Case Medical Center, University Hospitals Seidman Cancer Center, Case Comprehensive Cancer Center
Groups:
- Silicon Phthalocyanine 4 (0.1mg/ml) and PDT (50J/cm2): Level 1: Patients receive 0.1mg/ml silicon phthalocyanine 4 topically and then undergo 50J/cm2 PDT.
  silicon phthalocyanine 4: Given topically
  photodynamic therapy: Undergo PDT
  pharmacological study: Correlative studies
  laboratory biomarker analysis: Correlative studies
- Silicon Phthalocyanine 4 (0.1mg/ml) and PDT (100J/cm2): Level 2: Patients receive 0.1mg/ml silicon phthalocyanine 4 topically and then undergo 100J/cm2 PDT.
  silicon phthalocyanine 4: Given topically
  photodynamic therapy: Undergo PDT
  pharmacological study: Correlative studies
  laboratory biomarker analysis: Correlative studies
- Pc4 0.1(mg/ml) and Fluence 150(J/cm2): Level 3: Patients receive 0.1mg/ml silicon phthalocyanine 4 topically and then undergo 150J/cm2 PDT.
  silicon phthalocyanine 4: Given topically
  photodynamic therapy: Undergo PDT
  pharmacological study: Correlative studies
  laboratory biomarker analysis: Correlative studies
- Pc4 0.5(mg/ml) and Fluence 50(J/cm2): Level 4: Patients receive 0.5mg/ml silicon phthalocyanine 4 topically and then undergo 50J/cm2 PDT.
  silicon phthalocyanine 4: Given topically
  photodynamic therapy: Undergo PDT
  pharmacological study: Correlative studies
  laboratory biomarker analysis: Correlative studies
Period: Overall Study
Arm/Group | Silicon Phthalocyanine 4 (0.1mg/ml) and PDT (50J/cm2) | Silicon Phthalocyanine 4 (0.1mg/ml) and PDT (100J/cm2) | Pc4 0.1(mg/ml) and Fluence 150(J/cm2) | Pc4 0.5(mg/ml) and Fluence 50(J/cm2)
Started | 1 | 1 | 7 | 2
Completed | 1 | 1 | 7 | 2
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Silicon Phthalocyanine 4 (0.1mg/ml) and PDT (50 J/cm2): Patients receive 0.1mg/ml silicon phthalocyanine 4 topically and then undergo 50J/cm2 PDT.
  silicon phthalocyanine 4: Given topically
  photodynamic therapy: Undergo PDT
  pharmacological study: Correlative studies
  laboratory biomarker analysis: Correlative studies
- Silicon Phthalocyanine 4 (0.1mg/ml) and PDT (100 J/cm2): Patients receive 0.1mg/ml silicon phthalocyanine 4 topically and then undergo 100J/cm2 PDT.
  silicon phthalocyanine 4: Given topically
  photodynamic therapy: Undergo PDT
  pharmacological study: Correlative studies
  laboratory biomarker analysis: Correlative studies
- Silicon Phthalocyanine 4 (0.1mg/ml) and PDT (150 J/cm2): Patients receive 0.1mg/ml silicon phthalocyanine 4 topically and then undergo 150J/cm2 PDT.
  silicon phthalocyanine 4: Given topically
  photodynamic therapy: Undergo PDT
  pharmacological study: Correlative studies
  laboratory biomarker analysis: Correlative studies
- Silicon Phthalocyanine 4 (0.5mg/ml) and PDT (50 J/cm2): Patients receive 0.5mg/ml silicon phthalocyanine 4 topically and then undergo 50J/cm2 PDT.
  silicon phthalocyanine 4: Given topically
  photodynamic therapy: Undergo PDT
  pharmacological study: Correlative studies
  laboratory biomarker analysis: Correlative studies
- Total: Total of all reporting groups
Arm/Group | Silicon Phthalocyanine 4 (0.1mg/ml) and PDT (50 J/cm2) | Silicon Phthalocyanine 4 (0.1mg/ml) and PDT (100 J/cm2) | Silicon Phthalocyanine 4 (0.1mg/ml) and PDT (150 J/cm2) | Silicon Phthalocyanine 4 (0.5mg/ml) and PDT (50 J/cm2) | Total
Number analyzed (Participants) | 1 | 1 | 7 | 2 | 11
Age, Continuous [Median (Full Range); unit: years] | 63 [63 to 63] | 61 [61 to 61] | 51 [42 to 73] | 49 [41 to 57] | 55 [41 to 73]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 1 | 1 | 2
  Male | 1 | 1 | 6 | 1 | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 1 | 1 | 7 | 2 | 11
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 1 | 0 | 1
  White | 1 | 1 | 6 | 2 | 10
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 1 | 1 | 7 | 2 | 11
Fitzpatrick Skin Type Distribution [Number; unit: participants] — Type I (FST I): pale white skin, blue or hazel eyes, and blond or red hair who always burn and never tan. Type II (FST II): usually burn but can lightly tan with fair skin, blond or red hair, and blue, green or hazel eyes. Type III (FST III): sometimes mildly burn and develop a moderate tan. Type IV (FST IV): dark hair or brown eyes, who rarely burn and tan more than average. Type V (FST V): brown skin and have the same characteristics as FST IV. Type VI (FST VI): black skin and have the same characteristics as FST IV.
  participants
    FST I | 0 | 0 | 2 | 0 | 2
    FST II | 0 | 0 | 1 | 0 | 1
    FST III | 1 | 1 | 3 | 1 | 6
    FST IV | 0 | 0 | 1 | 1 | 2
    FST V | 0 | 0 | 0 | 0 | 0
    FST VI | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: MTD of Photodynamic Therapy
Description: Defined as the dose immediately below the dose in which 2 or more of 6 patients experience a grade 4 toxicity assessed using National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4.0.
Time Frame: Up to 30 days
Measure: Number; unit: J/cm^2
Arm/Group | Treatment (Silicon Phthalocyanine 4 and PDT)
Number analyzed (Participants) | 11
J/cm^2 | 150

2. Primary Outcome: MTD of Silicon Phthalocyanine 4 Defined as the Dose Immediately Below the Dose in Which 2 or More of 6 Patients Experience a Grade 4 Toxicity Assessed Using National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) Version 4.0
Time Frame: Up to 30 days
Measure: Number; unit: mg/ml
Arm/Group | Treatment (Silicon Phthalocyanine 4 and PDT)
Number analyzed (Participants) | 11
mg/ml | 0.1

ADVERSE EVENTS:
Time Frame: Patients will be followed for 30 days
Arm/Group | Treatment (Silicon Phthalocyanine 4 and PDT)
Serious Adverse Events (participants affected / at risk) | 0/11
Other Adverse Events (participants affected / at risk) | 11/11
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Silicon Phthalocyanine 4 and PDT) (N=11)
Peeling Skin (Skin and subcutaneous tissue disorders) | 1 (1)
Pain (Injury, poisoning and procedural complications) | 11 (29)
Cracked Tooth (Gastrointestinal disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1)
pruritus (Skin and subcutaneous tissue disorders) | 2 (2)
Sutures Removed (Injury, poisoning and procedural complications) | 1 (1)
Itching (Skin and subcutaneous tissue disorders) | 2 (2)
Elevated creatinine (Investigations) | 2 (2)
Hypertension (Vascular disorders) | 1 (1)
Palpitations (Cardiac disorders) | 1 (1)
Superficial ulceration (Skin and subcutaneous tissue disorders) | 2 (2)
Nose bleed (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sinusitis (Infections and infestations) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 1 (1)
Dermatitis (Injury, poisoning and procedural complications) | 1 (1)
excoriation (Skin and subcutaneous tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes